CLINICAL TRIAL: NCT06432530
Title: Can Hematological Inflammatory Indexes be Used to Differentiate Type 1 Modic Changes From Brucella Spondylodiscitis
Status: Completed | Type: Observational
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Volkan Şah, Principal Investigator, Yuzuncu Yil University
Other Study IDs: University of Van Yüzüncü Yıl
Record Dates: First submitted 2024-05-17; First posted 2024-05-29 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Brucella Spondylitis
MeSH Terms: interventions — C-Reactive Protein; Blood Sedimentation; Blood Cell Count

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 37 patients with type 1 Modic Changes (MCs): Diagnoses of brucella spondylodiscitis and type 1 MCs were supported by microbiological, serological, and radiological diagnostic tools. Based on the diagnostic tools and criteria, cases diagnosed with lumbar brucella spondylodiscitis or lumbar type 1 MCs in the past 5 years and who had simultaneously lumbar Magnetic Resonance Imaging (MRI), Complete Blood Count (CBC) test, C-reactive protein (CRP), and Erythrocyte Sedimentation Rate (ESR) results, and aged 18-65 years were selected to yield a study population
  Interventions: Other: C-Reactive Protein (CRP), Erythrocyte Sedimentation Rate (ESR), Complete Blood Count (CBC) values, and indexes derived from the CBC.
- 35 patients with brucella spondylodiscitis: Diagnoses of brucella spondylodiscitis and type 1 MCs were supported by microbiological, serological, and radiological diagnostic tools. Based on the diagnostic tools and criteria, cases diagnosed with lumbar brucella spondylodiscitis or lumbar type 1 MCs in the past 5 years and who had simultaneously lumbar Magnetic Resonance Imaging (MRI), Complete Blood Count (CBC) test, C-reactive protein (CRP), and Erythrocyte Sedimentation Rate (ESR) results, and aged 18-65 years were selected to yield a study population
  Interventions: Other: C-Reactive Protein (CRP), Erythrocyte Sedimentation Rate (ESR), Complete Blood Count (CBC) values, and indexes derived from the CBC.

INTERVENTIONS:
Other: C-Reactive Protein (CRP), Erythrocyte Sedimentation Rate (ESR), Complete Blood Count (CBC) values, and indexes derived from the CBC. — Patients' hematological parameters were recorded, and hematological inflammatory indexes (NLR: neutrophil/lymphocyte; MLR: monocyte/lymphocyte; PLR: platelet/lymphocyte; NLPR: neutrophil/(lymphocyte*platelet); SII (neutrophil*platelet/lymphocyte): systemic inflammatory index; SIRI (neutrophil*monocyte/lymphocyte): systemic inflammatory response index; AISI (neutrophil*platelet*monocyte/lymphocyte): aggregate index of systemic inflammation. ) were derived from baseline CBC tests.

SUMMARY:
Hematological inflammatory indices (Table 2) are currently very popular and have diagnostic, prognostic, and predictive, roles in various diseases. Considering their promising roles, we hypothesized that hematological inflammatory indices may have a distinctive value between brucella spondylodiscitis and type 1 Modic Changes (MCs). If the hypothesis is valid, early diagnosis-differential diagnosis-treatment processes may become easier and more successful. Given that hematological inflammatory indices are faster, practical, simpler, inexpensive, and easily accessible indicators, they may be more appropriate tools in differentiation between brucella spondylodiscitis and type 1 MCs.

DETAILED DESCRIPTION:
This is a retrospective comparative study focusing to distinguish between brucella spondylodiscitis and type 1 MCs considering hematological inflammatory indexes. Patients' data were obtained from Hospital Information Systems, between 2020 to 2024. A total of 35 patients with brucella spondylodiscitis and 37 type 1 MCs were enrolled in the study. Diagnoses of brucella spondylodiscitis and type 1 MCs were supported by microbiological, serological, and radiological diagnostic tools. Patients' hematological parameters were recorded, and hematological inflammatory indexes (NLR, MLR, PLR, NLPR, SII, SIRI, AISI) were derived from baseline CBC tests.

Based on the diagnostic tools and criteria1,2,14,21, cases diagnosed with lumbar brucella spondylodiscitis or lumbar type 1 MCs in the past 5 years and who had simultaneously lumbar MRI, Complete Blood Count (CBC) test, C-reactive protein (CRP), and erythrocyte sedimentation rate (ESR) results, and aged 18-65 years were selected to yield a study population. On the other hand, cases with inadequate data, aged <18 or >64 years, other infectious spondylodiscitis types than brucella, other MCs types than type 1, and other non-infectious conditions such as rheumatic spondylodiscitis (ankylosing spondylitis or Andersson lesion) were excluded from the study. Also, previous or recurrent brucella spondylodiscitis, involved other spinal levels than the lumbar spine were exclusion causes.

The two groups were statistically assessed and compared for baseline features such as age, gender, symptom duration, CRP, ESR, CBC values, and indexes derived from the CBC.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of lumbar brucella spondylodiscitis in the past 5 years
* Clinical diagnosis of or lumbar type 1 Modic Changes (MCs) in the past 5 years
* Having simultaneously lumbar Magnetic Resonance Imaging (MRI), Complete Blood Count (CBC) test, C-reactive protein (CRP), and erythrocyte sedimentation rate (ESR) results
* Being between the ages of 18-65

Exclusion Criteria:

* Cases with inadequate data
* Being under 18 years of age and over 65 years of age
* Having other infectious spondylodiscitis types than brucella
* Having other MCs types than type 1
* Having other non-infectious conditions such as rheumatic spondylodiscitis (ankylosing spondylitis or Andersson lesion)
* Having previous or recurrent brucella spondylodiscitis, involved other spinal levels than the lumbar spine

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: A total of 35 (17 female and 18 male) patients with brucella spondylodiscitis and 37 (26 female and 11 male) type 1 Modic Changes (MCs) were enrolled in the study. Diagnoses of brucella spondylodiscitis and type 1 MCs were supported by microbiological, serological, and radiological diagnotic tools. Patients' hematological parameters were recorded, and hematological inflammatory indexes (NLR: neutrophil/lymphocyte; MLR: monocyte/lymphocyte; PLR: platelet/lymphocyte; NLPR: neutrophil/(lymphocyte*platelet); SII (neutrophil*platelet/lymphocyte): systemic inflammatory index; SIRI (neutrophil*monocyte/lymphocyte): systemic inflammatory response index; AISI (neutrophil*platelet*monocyte/lymphocyte): aggregate index of systemic inflammation. ) were derived from baseline CBC tests.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2023-01-09 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2024-03-08 (Actual)

PRIMARY OUTCOMES:
C-Reactive Protein (CRP) | Baseline
  As an inflammatory index.
Erythrocyte Sedimentation Rate (ESR) | Baseline
  As an inflammatory index.
Neutrophil/Lymphocyte Rate (NLR) | Baseline
  As a hematological inflammatory index
Monocyte/Lymphocyte Rate (MLR) | Baseline
  As a hematological inflammatory index
Platelet/Lymphocyte Rate (PLR) | Baseline
  As a hematological inflammatory index
Neutrophil/(Lymphocyte*Platelet) Rate (NLPR) | Baseline
  As a hematological inflammatory index
(neutrophil*platelet/lymphocyte): Systemic Inflammatory Index (SII) | Baseline
  As a hematological inflammatory index
(neutrophil*monocyte/lymphocyte): Systemic Inflammatory Response Index (SIRI) | Baseline
  As a hematological inflammatory index
(neutrophil*platelet*monocyte/lymphocyte): Aggregate Index of Systemic Inflammation (AISI) | Baseline
  As a hematological inflammatory index

CONTACTS AND LOCATIONS:
Overall Officials: Ali İrfan Baran, Principal Investigator — Yüzüncü Yıl Üniversitesi Tıp Fakültesi
Locations (1):
- Volkan Şah, Van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No